CLINICAL TRIAL: NCT04529213
Title: Polygraphic Evaluation of the Effects of Different Rapid Maxillary Expansion Appliances on Sleep Quality: A Randomized Clinical Trial
Brief Title: Polygraphic Evaluation of the Effects of Different Rapid Maxillary Expansion Appliances on Sleep Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Gökçenur Gökçe, Assistant professor, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0024
Record Dates: First submitted 2020-08-24; First posted 2020-08-27 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Sleep Apnea Syndromes; Palatal Expansion Technique
Keywords: Polygraphy; Obstructive Sleep Apnea; Rapid Maxillary Expansion
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: 3-arm parallel trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tooth tissue-borne (KBME) expander (Experimental): In this tooth tissue-borne appliance, the occlusal surfaces of the molar and premolar teeth and half of the palatinal and buccal surfaces are covered with heat polymerized acrylic. Hyrax expansion screw is in the midline, as far as possible to the palate positioned close and parallel
  Interventions: Procedure: Rapid Maxillary Expansion Treatment
- Tooth-borne (Hyrax) expander (Experimental): In this tooth-borne expansion appliance, orthodontic bands are placed on the right and left 1st premolar and 1st molar teeth of the patients and the bands are soldered to the Hyrax expansion screw. The expansion screw is in the midline, as far as possible to the palate positioned close and parallel
  Interventions: Procedure: Rapid Maxillary Expansion Treatment
- Bone-borne (MIDME) expander (Experimental): This bone-borne expander includes 2 mini-screws with a diameter of 1.6 mm and a length of 10 mm on the right and left sides, coinciding between the roots of the 2nd premolar and 1st molar teeth in addition to the hyrax expansion screw.
  Interventions: Procedure: Rapid Maxillary Expansion Treatment

INTERVENTIONS:
Procedure: Rapid Maxillary Expansion Treatment — The patients were treated with KBME, Hyrax and MIDME maxillary expansion appliances, respectively. All expansion appliances containing a Hyrax expansion screw positioned parallel to the second premolars and were used to correct the posterior crossbite. In the MIDME group, two mini-screws with a diameter of 1.6 mm and a length of 10 mm are located on the right and left sides between the roots of the 2nd premolar and 1st molar teeth with 60-70° angle. KBME and Hyrax expansion appliances were cemented with glass ionomer cement and MIDME was cemented with using the light-cured composite. Same protocol was applied to all patients during RME treatment. Expansion screws in all groups were activated by two turns a day.

SUMMARY:
Rapid maxillary expansion (RME) is a commonly used orthodontic treatment in patients with maxillary constriction to provide skeletal expansion, correct posterior crossbite and resolve naso-respiratory problems by reducing oral respiration.The aim of this randomized controlled trial was to evaluate the effects of tooth-borne, tooth tissue-borne and bone-borne RME appliances on sleep quality with polygraphy. The null hypothesis was that there is no difference for the sleep quality between the appliances.

DETAILED DESCRIPTION:
Introduction. The aim of this 3-arm randomized controlled trial (RCT) was to evaluate the effects of tooth tissue-borne (KBME), tooth-borne (Hyrax), and bone-borne (MIDME) rapid maxillary expansion (RME) appliances on sleep quality with polygraphy.

Methods. This study was designed in parallel with an allocation ratio of 1:1:1. 46 patients with narrow maxilla and OSAS were included in this study and randomly assigned to three groups: tooth tissue-borne, tooth-borne and bone-borne expanders. Participants were congregated from the Department of Orthodontics, Faculty of Dentistry, Izmir Katip Celebi University, Turkey. In all groups, the expansion appliance was activated one-quarter turn twice a day until the desired suture opening was achieved. The primary outcome of this study was the correction of posterior crossbite. Secondary outcomes included polygraphic assessment of sleep parameters. Each subject participated in 1 overnight sleep test with polygraphy before the expansion (T0) and after a 3-month retention phase of treatment (T1). According to the results of polygraphy, 7 parameters; (apnea hypopnea index (AHI), number of apnea and hypopnea, desaturation index, lowest desaturation, average saturation, supin AHI) were examined to evaluate the changes in sleep scores. Kruskal-Wallis analysis and Dunn-Bonferroni test were used for inter-group comparisons and Wilcoxon analysis was used for intra-group evalaution. P<0.05 was accepted statistically significant. Computer-generated randomization was used with group allocation concealed using opaque, sealed envelopes. The outcome assessor was blinded to group assignment. The outcome assessor was blinded; however, it was not feasible to blind either operator or patients.

ELIGIBILITY:
Inclusion Criteria:

1. No previous tonsillar, nasal or adenoid surgery and orthodontic treatment,
2. Bilateral crossbite and need for RME,
3. Maxillary and mandibular permanent teeth fully erupted,
4. Willingness to participate in the study

Exclusion Criteria:

1. the presence of adenotonsillectomy due to tonsillar hypertrophy or adenoidal hypertrophy
2. having nasal/nasopharyngeal /oropharyngeal pathologies, craniofacial syndromes, systemic disease, poor oral hygiene,
3. history of previous orthodontic treatment.

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-01-13 (Actual); Study Completion 2017-05-17 (Actual)

PRIMARY OUTCOMES:
Correction of posterior crossbite | After active expansion (up to 3 weeks). The evaluation of the result has been made by the physician with intraoral clinical examination.
  The palatal cusps of the maxillary posterior teeth approximated the lingual cusps of the mandibular posterior teeth.

SECONDARY OUTCOMES:
Polygraphic assessment of sleep parameters | After 3 months treatment retention period
  Changes in apnea hypopnea index (AHI)
Polygraphic assessment of sleep parameters | After 3 months treatment retention period
  Changes in number of apnea and hypopnea
Polygraphic assessment of sleep parameters | After 3 months treatment retention period
  Changes in number of hypopnea
Polygraphic assessment of sleep parameters | After 3 months treatment retention period
  Changes in desaturation index
Polygraphic assessment of sleep parameters | After 3 months treatment retention period
  Changes in lowest desaturation
Polygraphic assessment of sleep parameters | After 3 months treatment retention period
  Changes in average saturation
Polygraphic assessment of sleep parameters | After 3 months treatment retention period
  Changes in the value of Supin AHI

CONTACTS AND LOCATIONS:
Overall Officials: Gökçenur Gökçe, Phd, Principal Investigator — Izmir Katip Celebi University

IPD SHARING:
Plan to Share IPD: Undecided